CLINICAL TRIAL: NCT00959907
Title: A Phase iv Controlled Randomized Blinded Study on the Anhydrotic Action Halos and Muscle Activity of Two Commercial Preparations Type a Botulinum Toxin (Dysport® and Botox® ) Administered to the Upper Third of the Face
Brief Title: Comparison of Two Commercial Preparations of Botulinum Toxin Type A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hexsel Dermatology Clinic (Other)
Responsible Party: Doris Hexsel, CBED
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-CBED06
Record Dates: First submitted 2009-04-23; First posted 2009-08-17 (Estimated); Results first posted 2009-08-17 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-11

CONDITIONS: Wrinkles in Frontal Area
Keywords: Muscular activity; wrinkles in frontal area; action halos
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BoNT A1 (4U) (Active Comparator): BoNT A1 (4U): Botulinum toxin A (Dysport®)4 units
  Interventions: Drug: BOTULINUM TOXIN TYPE-A
- BoNT-A2 (2U) (Active Comparator): BoNT-A2(2U): Botulinum toxin A (Botox®) 2 units
  Interventions: Drug: BOTULINUM TOXIN TYPE-A

INTERVENTIONS:
Drug: BOTULINUM TOXIN TYPE-A — On Visit 1 (Day 0):
  Botulinum toxin A (Dysport® and Botox®) will be administered according to an equivalence ratio of 2:1. Both reconstituted in the same volume per point, injected in the forehead determined site.
  * Dysport®: 4 units will be injected in the left or right forehead side.
  * Botox® : 2 units will be injected in the left or right forehead side.(opposite side of dysport injection)
  Other Names: BoNT A1 = Dysport; BoNT A2 = Botox

SUMMARY:
The objective of this study is to compare the action halos of the botulinum toxins (Dysport® and Botox®) using two equivalence-ratios and to gather supportive information, such as more detailed data on the effectiveness in reduction of wrinkles and duration of action on the upper part of the face of both products, trough scales and photographs evaluations.

DETAILED DESCRIPTION:
This was a monocentric, prospective, randomized and double-blind study. Fifty nine female patients, presenting with moderate to severe forehead wrinkles, with sweating ability who had never undergone previous BoNT-A injections were enrolled. There were two randomizations, one related to the dose-equivalence (2:1U and 2.5:1U), both reconstituted in the same volume of 0.02 mL per point and another related to the forehead side (left or right) for application of the tested drugs. Baseline, twenty-eight and 112 days later, clinical and photographic assessments, Minor´s test, and electromyographic (EMG) evaluations were performed.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent (Annex 1)
2. Female
3. Subjects agreeing to take part in all procedures of the study, including botulinum toxin applications, Minor's test, measurement of Evoked Potentials, photographs, etc.), after being fully informed on the objectives and nature of the investigations
4. Subjects aged between 18 and 60 years
5. Subjects presenting with moderate to severe wrinkles on the forehead under maximum voluntary contraction of the m. frontalis
6. Subjects with positive Minor's test showing sweating on the forehead in standardized conditions described in Annex 2

   *The Minor's Test will be the last inclusion criterion to be evaluated. Only these patients eligible according to the other inclusion criteria will undergo the Minor's Test to evaluate their sweating on the forehead. The cut off point is a positive Minor's Test (Level +1) - only subjects with Minor's Test (Level +1) will be recruited in the study (Annex 2).
7. Medical history and physical examination which, based on the investigator's opinion, do not prevent the patient from taking part in the study and use the products under investigation
8. Subjects of childbearing age should present a negative urine pregnancy test at baseline and should be using an effective contraceptive method;
9. Availability of the patient throughout the duration of the study (112 days)
10. Subject agrees not to undergo other cosmetic or dermatological procedures during the study
11. Subjects with sufficient schooling and awareness to enable them to cooperate to the degree required by this protocol

Exclusion Criteria:

1. Pregnant women or women intending to become pregnant in the next 4 months after screening for eligibility
2. Subjects who are lactating
3. Subjects having undergone botulinum toxin treatment within the last 6 months
4. Subjects participating in other clinical trials
5. Any prior surgery affecting the frontalis and/or orbicularis muscles, prior blepharoplasty or brow lift
6. Any prior cosmetic procedures, including fillers, or scars that may interfere with the study results
7. Subjects presenting fronto-parietal alopecia according to the Norwood-Hamilton classification
8. Subjects with neoplastic, muscular or neurological diseases
9. Subjects using aminoglycoside and penicillamine antibiotics, quinine and Ca2+ channel blockers
10. Subjects with inflammation or active infection in the area to be injected
11. Subjects presenting evident facial asymmetry
12. Subjects with a history of adverse effects, such as sensitivity to the components of the formula, ptosis or any other adverse effect, which in the investigator's opinion should prevent the patient from participating in the study
13. Subjects presenting myasthenia gravis, Eaton-Lambert Syndrome and motor neuron diseases
14. Subjects with coagulation disorders or using anticoagulants
15. Subjects with known systemic autoimmune diseases
16. Subjects with a history of medical treatment non-adherence or showing unwillingness to adhere to the study protocol
17. Any condition that, in the opinion of the investigator, can compromise the evaluation of the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2005-05; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris Hexsel, MD, Principal Investigator
Locations (1):
- Brazilian Center for Dermatological Studies, Porto Alegre, Rio Grande do Sul, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment process: It is planned to recruit a total of 58 subjects at one single centre, Brazilian Center For Studies in Dermatology, in Porto Alegre, Brazil. The anticipated drop out rate is 10%.
  Baseline evaluation: May 2005 to July 2007.
Pre-assignment Details: 13 volunteers were excluded; (screen failure) Iodine allergy=2 Minor´s Test failure=6 Mild wrinkles=3 Inclusion criteria failure=2
Groups:
- BoNT A1(4U): Group 1: Botulinum toxin A (Dysport®) will be administered 4 units of Dysport®
- BoNT-A2(2U): Group 2: Botulinum toxin A (Botox®) will be administered 2 units of Botox®
Period: Overall Study
Arm/Group | BoNT A1(4U) | BoNT-A2(2U)
Started | 30 | 29
Completed | 27 | 28
Not Completed | 3 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BoNT A1(4U) | BoNT-A2(2U) | Total
Number analyzed (Participants) | 30 | 29 | 59
Age Continuous [Mean (Standard Deviation); unit: years] | 44.77 (8.67) | 41.86 (11.98) | 42.88 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 59
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Horizontal Action Halo Diameter at 28 Days
Description: Minor's test permits the visualization of the effect of botulinum toxin in the injected area,also called action halos. Mirror is a computer program that allows, through photogrpahs, measuring the horizontal diameter and the area of action halos.
Time Frame: 28 days
Population: The analysis was intention to treat (ITT); One drop out, from baseline to visit 1(intervention) and 3 drop outs from visit 1 to visit 2 (28 days after botulinum toxin injections). Started 59 volunteers - 4 drop outs, there was 55 volunteers in the first analysis.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | BoNT A1(4U) | BoNT-A2(2U)
Number analyzed (Participants) | 27 | 28
centimeter | 1.0526 (0.3638) | 1.0670 (0.2239)
Statistical Analysis 1: Comparison: BoNT A1(4U); Test type: Superiority or Other; p = 0.832, t-test, 2 sided

2. Primary Outcome: ECMAP in m. Frontialis BoNT A1(4U) X BoNT A2 (2U)
Description: ECMAP(Evoked Compound Muscle Action Potentials) was accessed by an electromyography (EMG) device (TECA Sapphire - TECA Corp., Pleasantville, NY).
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | BoNT A1(4U) | BoNT-A2(2U)
Number analyzed (Participants) | 28 | 28
microvolts | 276.18 (319.15) | 289.00 (303.86)
Statistical Analysis 1: Comparison: BoNT A1(4U); Test type: Superiority or Other; p = 0.658, t-test, 2 sided
Statistical Analysis 2: Comparison: BoNT-A2(2U); Test type: Superiority or Other; p = 0.739, t-test, 2 sided

3. Primary Outcome: Horizontal Action Halo Diameter at 112 Days
Description: as for outcome 1
Time Frame: 112 days
Population: Intention to treat analysis. 55 volunteers - One drop out from visit 2 (28 days) to visit 3 (112 days): 54 volunteers.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | BoNT A1(4U) | BoNT-A2(2U)
Number analyzed (Participants) | 26 | 28
centimeter | 0.8742 (0.3333) | 1.1196 (0.2620)
Statistical Analysis 1: Comparison: BoNT A1(4U); Test type: Superiority or Other; p = 0.184, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | BoNT A1(4U) | BoNT-A2(2U)
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

LIMITATIONS AND CAVEATS:
The field of muscular effects of the studied toxins was objectively measured by EMG and it is not very precise. However, there is no more precise objective measurement to currently evaluate the field effects in muscles than EMG.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No